CLINICAL TRIAL: NCT03988790
Title: Evaluation of Response to Monoclonal Antibody Therapy in Severe Asthma: Research of Predictive Biomarkers in Exhaled Air
Brief Title: Evaluation of the Response to Monoclonal Antibody Therapy in Severe Asthma: Research of Predictive Biomarkers in Exhaled Air
Acronym: Zina-VOC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018_0075
Record Dates: First submitted 2019-06-06; First posted 2019-06-17 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Single Group Assignement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VOC analysis (Experimental): VOC analysis in exhaled air in patients with severe asthma treated by monoclonal antibody
  Interventions: Device: VOC analysis

INTERVENTIONS:
Device: VOC analysis — VOC analysis in exhaled air with e-noses and mass spectrometry.

SUMMARY:
This study evaluates the change in the composition of Volatil Organic Compounds (VOC) in patients treated by monoclonal antibody for severe asthma.

DETAILED DESCRIPTION:
At least one in two patients treated by monoclonal antibody for severe asthma doesn't have satisfying result after 6 months of treatment.

The evaluation of the answer, and even better the answer prediction, are fundamental issues for medico-economic plan as part of these innovative therapeutics.

The interest of the use of VOC as diagnostic or prognostic tool in patients with tumoral thoracic pathology or bronchial or pulmonary vascular diseases has been demonstrated.

VOC analysis will be performed using two different techniques: electronic nose and masse spectrometry. At each visit, in addition to the usual assessment, patients will have two non-invasives collections of exhaled air, one for electronic nose analysis and one for masse spectrometry analysis.

ELIGIBILITY:
Inclusion Criteria:

* patient aged > 18 years old
* patient with severe asthma who respond to the indication of monoclonal antibody therapy according to SPC and management criteria fixed by Transparency Committee
* signed informed consent
* patient with healthcare insurance

Exclusion Criteria:

* patient not responding to the criteria for the good use of monoclonal antibody in severe asthma
* contraindication to one of monoclonal antibody treatment according to SPC (hypersensitivity to one of compounds)
* patient unable to perform a slow vital capacity
* patient with long-term oxygen therapy , under invasive ventilation
* pregnant women
* patient deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-12-04 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Volatil Organic Compound (VOC) profiles predictive of clinically significant response | 1 day
  Clinically significant response defined by:
  * reduction of 50% of number of exacerbations treated by oral corticosteroids after 12 months of treatment compared to the number of exacerbation during the previous year AND/OR
  * increase of 3 points (MCID according to Schartz and al 2009) of ACT score after 3 months of treatment and maintained at 6 months

SECONDARY OUTCOMES:
Change of FEV and FEV/CV | change from baseline profiles at 3, 6 and12 months post-baseline
  Predictive variations of a clinically relevant response with improvement of FEV and FEV/CV at 3, 6 and 12 months
Decrease of residual volume | change from baseline profiles at 3, 6 and12 months post-baseline
  Predictive variations of a clinically relevant response with decrease of residual volume (RV) at 3, 6 and 12 months
Decrease of the daily dose of oral corticosteroids | change from baseline profiles at 1, 3, 6 and12 months post-baseline
  Predictive variations of a clinically relevant response with decrease of the daily dose of oral corticosteroids for corticosteroid-dependent patients at 1, 3, 6 and 12 months
Reduction in the number of exacerbations | change from baseline profiles at 1, 3, 6 and12 months post-baseline
  50% reduction in the number of exacerbations treated with oral steroids after 6 months of treatment compared to the number of exacerbations in the previous year OR a 3 point increase in the ACT (Asthma Control Test) score after 3 months of treatment maintained at 6 months OR increase of GETE (global evaluation of treatment effectiveness) score at 1, 3, 6 and 12 months
Change before and after treatment | change from baseline profiles at 12 months post-baseline
  Change of Volatil Organic Compound (VOC) profiles before and after treatment whatever is the clinical answer
Change according to administered antibody | 1 day
  Change of Volatil Organic Compound (VOC) profiles according to administered antibody
Volatil Organic Compound (VOC) profiles according to patients' phenotype | 1 day
  Volatil Organic Compound (VOC) profiles according to patients' phenotype at the inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Devillier, Principal Investigator — Pneumology department
Locations (1):
- Hôpital Foch, Suresnes, France